CLINICAL TRIAL: NCT02343770
Title: Usefulness of Protoarray®Microarray for Identifying Biomarkers in Idiopathic Juvenile Arthritis Antinuclear Antibodies Positive.
Brief Title: Biomarkers in Idiopathic Juvenile Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9355
Record Dates: First submitted 2015-01-07; First posted 2015-01-22 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Idiopathic Juvenile Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- idiopathic juvenile arthritis (Experimental): blood sample
  Interventions: Other: blood sample for identifying biomarkers
- control (Other): blood sample
  Interventions: Other: blood sample for identifying biomarkers

INTERVENTIONS:
Other: blood sample for identifying biomarkers

SUMMARY:
Juvenile idiopathic arthritis (JIA) is the most common form of arthritis in children. The etiology is unknown. Several types of arthritis fall under the JIA heading. Oligoarticular JIA with antinuclear antibodies affects about half of all children. There 's no specific markers. Our purpose is to identify new markers in this pathology. The ProtoArray®Human Protein Microarray allows rapid and efficient detection of protein interaction using a suitable protein or small molecule probe. The investigators hope so detect novel potential autoantigen biomarkers specific in JIA.

DETAILED DESCRIPTION:
We select 10 patients with inclusion criteria and 10 controls. We analyse their blood sample (5ml). The ProtoArray® Microarray allows to detect novel protein-protein interactions, to rapidly perform serum profiling using a sensitive method to detect potential autoantigen biomarkers. The ProtoArray® Human Protein Microarray is a high-density protein microarray containing thousands of purified human proteins for protein interaction screening.

ELIGIBILITY:
Inclusion Criteria for experimental group :

* child age from 2 to 16 years
* Oligoarticular JIA with antinuclear antibodies
* with or without uveitis

Exclusion criteria for experimental group :

* immunosuppressive and biological therapy

Inclusion Criteria for control group :

* child age from 2 to 16 years

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
identification of specific autoantigen biomarkers | 1 day
  Identify blood sampling biomarkers of juvenile idiopathic arthritis

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology paediatric consultation, Arnaud de Villeneuve Hospital, Montpellier, France